CLINICAL TRIAL: NCT04941053
Title: Seroprevalence of COVID19 in Sohag Governorate Egypt
Brief Title: Seroprevalence of COVID-19
Acronym: cov prevalence
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Saber Shafik, lecturer, Sohag University
Other Study IDs: Soh-Med-21-04-33
Record Dates: First submitted 2021-06-23; First posted 2021-06-28 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1 chronic haemodialysis patients: seroprevalnce of COVID 19
  Interventions: Diagnostic Test: laboratory test
- healthy control: seroprevalnce of COVID 19
  Interventions: Diagnostic Test: laboratory test

INTERVENTIONS:
Diagnostic Test: laboratory test — seroprevalnce

SUMMARY:
Coronavirus disease pandemic has been started in late 2019. Since this date, the number of cases has been increased reaching 32.7 million cases worldwide in 27 September, 2020. . Herd immunity is achieved when enough people become immune to a virus to stop its spread. Around 70% to 90% of a population needs to be immune to protect the uninfected. In A Spanish study of more than 30,000 people estimates that around just 5% of the Spanish population has developed antibodies

DETAILED DESCRIPTION:
Aims of work:

A cross-sectional study to detect the seroprevalence to COVID 19 in chronic hemodialysis patients and compare it with the COVID 19 seroprevalence in healthy control in Sohag governorate Egypt

Methods:

After taken informed consent according to Sohag University Ethical Committee A questionnaire on coronavirus symptoms will be asked including epidemiological characters and history of previous COVID 19 infection and infection control measures to prevent it

5 ml of the blood sample will be taken for IgG antibodies testing with a chemiluminescent microparticle immunoassay.

ELIGIBILITY:
Inclusion Criteria:

* patient accept to participate

Exclusion Criteria:

* vaccinated people

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: group 1 patients coming to hemodialysis unit group 2 relative to patients coming to hemodialysis unit, medical staff
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
seroprevalnce | 3-6-2021 to 30-8-2021
  antibody measurement

CONTACTS AND LOCATIONS:
Overall Officials: N S shafik, lecturer, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
to protect privacy of data of patients